CLINICAL TRIAL: NCT05946291
Title: The Effect of Two Different Simulation Applications on the Level of Pressure Injury Knowledge and Evaluation in Nursing Students: A Randomized Controlled Trial
Brief Title: Simulation Applications on the Level of Pressure Injury Knowledge and Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Zilan BARAN, Principal Investigator, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TepecikTRH NURSE
Record Dates: First submitted 2023-05-17; First posted 2023-07-14 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Pressure Injury
Keywords: pressure injury; nursing students; simulation; moulage
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The study is planned as a double-blind randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Students will be assigned to the experiment and control group blind. In addition, double-blind randomization will be provided by appointing a blind researcher who performs the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Patient Group (Experimental): Standardized Patient: A pressure wound similar to reality will be created with the application of mulage on a standardized patient. In accordance with the scenario of a patient with a pressure wound, students will perform pressure wound evaluation and maintenance on a standardized patient in a simulation laboratory. Following the simulation application, student groups of eight to ten individuals will participate in a debriefing session.
  Interventions: Other: Pressure injury training
- Simulated Manneqquin Group (Active Comparator): Simulated Mannequin: A pressure wound similar to reality will be created with the simulated mannequin mulage application. In accordance with the same scenario used in the experimental group, pressure wound evaluation and maintenance will be performed on the simulated mannequin in the simulation laboratory. Following the simulation application, student groups of eight to ten individuals will participate in a debriefing session.
  Interventions: Other: Simulated Manneqquin training

INTERVENTIONS:
Other: Pressure injury training — Pressure injury training with mulage application on a standardized patient
  Arms: Standardized Patient Group
Other: Simulated Manneqquin training — Pressure injury training with mulage application on a simulated manneqquin
  Arms: Simulated Manneqquin Group

SUMMARY:
When the literature is examined, it is seen that the pressure injury knowledge and evaluation levels of nursing students are low. Today, innovative approaches have started to be introduced to nursing education in proportion to the development of technology. Simulation applications are also seen as one of these innovative approaches. In our study, it is aimed to examine the effect of pressure injury training to be given using high-reality standardized patient use and a medium-reality simulation model on the knowledge and evaluation level of intern nursing students. Students (n = 250) will be assigned blindly to the experimental and control groups using a simple randomization method, and then pressure injury information and assessment trainings will be given to the experimental group with a medium-reality simulation model on a standardized patient for the control group for 4 weeks. After 2 weeks, the final test will be performed, and the data will be assigned to blind groups. It will be evaluated by the researcher.

DETAILED DESCRIPTION:
According to the literature, it is seen that nursing students do not have sufficient knowledge about pressure injuries, and innovative applications are needed to improve their clinical skills. When the studies are examined, it is seen that the studies comparing standardized patient use and simulation application in pressure injury education for nursing students are very limited. In this context, it is seen that there is a need for studies in which the effectiveness of different simulation applications in learning pressure injury in nursing students is examined, and it is considered important to contribute to the literature with this study to be conducted. It is considered that the project has the potential to be published in internationally respected journals and presented at conferences. Due to the increase in the number of students in nursing education and the lack of clinical areas, it is extremely important to practice in reality-like environments. In addition, students are required to acquire nursing psychomotor skills before meeting with a real patient. In this study, it is aimed to examine the effect of pressure injury teaching performed with standardized patients and a medium-reality simulation model on the knowledge and evaluation levels of nursing students. In this context, the hypothesis of the study is:

H0: There is no difference between the knowledge and evaluation levels of pressure injury in nursing students of the teaching given using standardized patient and medium-reality simulation model applications. H1: There is a difference between the knowledge and evaluation levels of pressure injury in nursing students based on the teaching given using standardized patient and medium-reality simulation model applications. In this study, it is planned to provide two different types of simulation training aimed at improving the knowledge and evaluation levels of nursing students about pressure injuries. The use of simulation applications will increase the psychomotor skills of the student and increase the level of knowledge and evaluation without encountering the real patient. In addition, the standardized patient and medium-reality simulation model planned to be used in the study will provide many students with the opportunity to learn about pressure injuries without the need to train on patients in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Intern nursing students

Exclusion Criteria:

* Students who have previously received Care Management lecture or wound care training
* Have come with a horizontal transfer
* Have graduated from health vocational high school
* Work in a hospital or other institution
* Do not volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
As a result of the study, it is expected that there will be an change in the students' pressure injury knowledge level. | Before and two weeks following applications
  The Turkish version of the Pressure Ulcer Knowledge Assessment Tool-updated version (PUKAT 2.0)" was developed in 2022 as a tool to assess the level of knowledge of pressure ulcers among nurses. It is a 25-question measurement tool consisting of a total of 6 sub-dimensions, including etiology of pressure injury, classification and observation, risk assessment, nutrition, prevention of occurrence, and special patient groups, with 5 Likert-type options. It was reported to have valid and reliable psychometric properties, as indicated by a Cronbach's Alpha value of 0.72, and to be suitable for use in the evaluation of the level of knowledge regarding pressure injuries. The minimum and maximum values obtainable from the scale are 0 and 25, respectively. The higher the score, the higher the level of knowledge.
As a result of the study, it is expected that there will be an change in the level of pressure injury assessment of students. | Before and two weeks following applications
  The Pressure Injury Staging Registration Form was developed by the researchers. This form consists of pressure injuries at different stages, a total of 25 of which were taken by a wound care nurse. The form and photos have been submitted to three expert suggestions and have taken their final shape in accordance with the suggestions received. 5 of the photos include stage 1, 5 of them stage 2, 5 of them stage 3, 5 of them stage 4, 3 of them are non-staged pressure injuries, and 2 of them are deep tissue injuries.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dalli OE, Yildirim Y, Caliskan G, Girgin NK. Reliability and validity of the Turkish version of pressure ulcer knowledge assessment tool-updated version (PUKAT 2.0). J Tissue Viability. 2022 Feb;31(1):52-57. doi: 10.1016/j.jtv.2021.08.001. Epub 2021 Aug 11. PMID 34429220
- [Derived] Baran Z, Ayik C, Ozden D. Comparison of standardized patient and medium-fidelity simulation practices on nursing students' knowledge, staging, and satisfaction regarding pressure injuries: A randomized controlled trial. Nurse Educ Today. 2025 Aug;151:106735. doi: 10.1016/j.nedt.2025.106735. Epub 2025 Apr 2. PMID 40209560